CLINICAL TRIAL: NCT02488512
Title: Peptide Receptor Radionuclide Therapy With 90Y-Dotatoc in Relapsed/Refractory Diffuse Large B Cell (DLBCL) and Mantle Cell Lymphomas (MCL)
Brief Title: Peptide Receptor Radionuclide Therapy With 90Y-Dotatoc in Relapsed/Refractory Diffuse Large B Cell and Mantle Cell Lymphomas
Acronym: itTRIOlym
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: critical low recruitment rate
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST202.02
Record Dates: First submitted 2015-06-19; First posted 2015-07-02 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: DLBCL; MCL; Recurrent Disease
Keywords: Relapsed/refractory diffuse large b cell; Relapsed/refractory mantle cell lymphomas; DLBCL; MCL; 90Y-DOTATOC; SSR-positive tumour
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell | interventions — 90Y-octreotide, DOTA-Tyr(3)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 90Y-DOTATOC (Experimental): 90Y-DOTATOC
  Interventions: Drug: 90Y-DOTATOC

INTERVENTIONS:
Drug: 90Y-DOTATOC — Each patient will receive a maximum cumulative 90Y-DOTATOC activity of 11.1 GBq (300 mCi) [45-46], divided into 4 cycles (1.8 - 2.8 GBq for each cycle) with an interval of 6 - 8 weeks between cycles. The activity to be administered will be measured in a dose calibrator, properly calibrated for the 90Y-radionuclide.
  Other Names: Y-PRRT

SUMMARY:
This is a prospective, single arm,single centre open-label, phase II study in relapsed or refractory DLBCL and MCL non-Hodgkin's lymphoma (NHL), not suitable to other therapies, included HDCT, or patients relapsed after high-dose chemotherapy (HDCT) with autologous stem-cell transplantation (ASCT), treated with peptide receptor radionuclide therapy with 90Y-Dotatoc.

Each patient will receive a maximum cumulative 90Y-DOTATOC activity of 11.1 GBq (300 mCi), divided into 4 cycles (1.8 - 2.8 gigabequerel (GBq) for each cycle) with an interval of 6 - 8 weeks between cycles. The 90Y-DOTATOC will be slowly infused intravenously.

35 patients will be enrolled in 36 months in two stages (18 patients in the first stage, if 2 or fewer patients will show an objective response, the study will be closed).

DETAILED DESCRIPTION:
PEPTIDE RECEPTOR RADIONUCLIDE THERAPY (PRRT) WITH 90Y-DOTATOC IN RELAPSED/REFRACTORY DIFFUSE LARGE B CELL AND MANTLE CELL LYMPHOMAS.

This is a prospective, single arm, open-label, phase II study. It is estimated that a maximum of 35 patients will be enrolled in 36 months; the treatment efficacy will be tested in 18 patients in the first stage, if 2 or fewer patients will show an objective response, the study will be closed; if > 2 objective responses will be observed, a total of 35 patients will be enrolled.

Follow up period is 48 months.

Single-center

The primary objective is the evaluation of objective response rate (ORR). of Y-PRRT in relapsed or refractory DLBCl and MCL NHL, not suitable to other therapies, included HDCT, or patients relapsed after HDCT with ASCT.

The secondary objectives are toxicity (acute and late), progression free survival, overall survival and Quality of life.

35 patients will be enrolled in 36 months in two stages (18 patients in the first stage, if 2 or fewer patients will show an objective response, the study will be closed).

Each patient will receive a maximum cumulative 90Y-DOTATOC activity of 11.1 GBq (300 mCi), divided into 4 cycles (1.8 - 2.8 GBq for each cycle) with an interval of 6 - 8 weeks between cycles. The 90Y-DOTATOC will be slowly infused intravenously.

The study will be conducted following the Optimal Two Stage Design assuming the true response probability:

* under H0 (p0) <=10%
* under H1 (p1) >=30% and considering alpha=0.05 and power=0.90.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged >18 years.
2. Histologically confirmed relapsed or refractory DLBCL or MCL not suitable to other treatments.
3. Patients with documented disease will be admitted to therapeutic phase only if the diagnostic PET/CT with 68Ga-DOTATOC images demonstrate a significant uptake in the tumour (SSR-positive tumour).
4. Patients must have at least one bidimensional measurable lesion with long axis > 15 mm at CT scan (MRI is allowed only if CT scan cannot be performed), according to Cheson Criteria.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Life expectancy of at least 3 months.
7. Adequate cardiac function as assessed at echocardiography and ECG.
8. Conserved hematological, liver and renal parameters, and in particular: haemoglobin >= 9 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X UNL (upper normal limit), Alanine aminotransferase (ALT) <2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL
9. Patients must not have received other treatments with radiopeptides (e.g. 111In-pentetreotide, 177Lu-DOTATATE, 131I-MIBG).
10. If female of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at screening visit and continuing until 3 months following last treatment with study drug. Negative serum pregnancy test for females of childbearing potential within 7 days of starting treatment.

Exclusion Criteria:

1. Pregnancy/breastfeeding (a pregnancy test not older than 7 days is mandatory).
2. Bone marrow invasion > 25 %.
3. Other concomitant neoplasm (excluding in situ basaliomas and radically treated cervical cancers); subjects must be free from other neoplasms at least 3 years. All acute toxic effects of any prior therapy (including surgery radiation therapy,chemotherapy) must have resolved to a grade <= 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE).
4. Evidence of myelodysplastic syndrome or other hematologic diseases
5. Patients treated with chemotherapy and therapeutic radiotherapy within 4 weeks.
6. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Positive serology for Hepatitis B (HB) defined as a positive test for Hepatitis B surface antigen (HbsAg). In addition, if negative for HBsAg but Hepatitis B core antibody (HBcAb) positive (regardless of HBsAb status), a hepatitis B virus (HBV) DNA test will be performed and if positive the subject will be excluded. Any patient with HBcAb positivity will receive anti viral prophylaxis during the study, according to the procedures suggested by local Hepatology service.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition.
10. Previous autologous stem cell transplant in the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
overall response rate (ORR) | up to 48 months
  ORR will be calculated according to Response Evaluation Criteria in Non Hodgkin's lymphoma according to Cheson Criteria

SECONDARY OUTCOMES:
acute toxicity evaluation | up to 48 months
  The acute toxicity will be recorded according to the CTC-AE, version 4.0 in the safety population until Follow-up is completed (48 months).
progression free survival (PFS) | up to 48 months
  PFS is defined as the time from the start treatment date to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation
overall survival (OS) | up to 48 months
  OS is defined as the time from treatment start to the time of death from any cause. Subjects who are alive at the time of the final analysis or who have become lost to follow-up will be censored at their last known alive date.
Quality of Life (QLQ) | up to 48 months
  Quality of life will be evaluated with Version 3.0 European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
late toxicity evaluation | up to 48 months
  The late toxicity will be recorded according to the CTC-AE, version 4.0 in the safety population until Follow-up is completed (48 months) .

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (1):
- Nuclear Medicin Division, IRST IRCCS, Meldola, FC, Italy